CLINICAL TRIAL: NCT00742625
Title: Dose Escalation and Phase II Study of Bortezomib (IND #58443) Added to Standard Daunorubicin and Cytarabine Therapy for Patients With Previously Untreated Acute Myeloid Leukemia Age 60-75 Years
Brief Title: Bortezomib, Daunorubicin, and Cytarabine in Treating Older Patients With Previously Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00443; NCI-2009-00443 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000612758; CALGB 10502 (Other: Cancer and Leukemia Group B); CALGB-10502 (Other: CTEP); U10CA031946 (NIH); P30CA014236 (NIH); NCT01647061 (obsolete NCT alias)
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-06

CONDITIONS: Acute Myeloid Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Daunorubicin; Cytarabine; Bortezomib

ARMS (1):
- Treatment (daunorubicin hydrochloride and bortezomib) (Experimental): See Detailed Description
  Interventions: Drug: daunorubicin hydrochloride; Drug: cytarabine; Drug: bortezomib

INTERVENTIONS:
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
This phase II trial studies the side effects and best dose of bortezomib when given together with daunorubicin and cytarabine and to see how well it works in treating older patients with previously untreated acute myeloid leukemia. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as daunorubicin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the remission induction response rate (complete response [CR] and CR with incomplete platelet recovery [CRp]) in older patients with previously untreated acute myeloid leukemia treated with induction therapy comprising bortezomib in combination with daunorubicin hydrochloride and cytarabine.

II. To define the maximum tolerated dose of bortezomib when administered in combination with intermediate-dose cytarabine after induction therapy.

SECONDARY OBJECTIVES:

I. To describe the disease-free survival of patients treated with this regimen. II. To describe the overall survival of patients treated with this regimen. III. To evaluate the treatment-related toxicities in these patients.

OUTLINE: This is a multicenter, dose-escalation study of bortezomib. Doses of bortezomib are escalated during remission consolidation therapy.

REMISSION INDUCTION THERAPY: Remission induction course 1: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11; daunorubicin hydrochloride IV on days 1-3; and cytarabine IV continuously over 168 hours on days 1-7.

After completion of remission induction course 1, patients undergo bone marrow aspiration and biopsy for evaluation of response. Patients achieving a complete response (CR) or partial response (PR) proceed to remission consolidation therapy. Patients achieving a CR with incomplete platelet recovery (CRp) proceed to remission consolidation therapy after platelet counts recover. Patients with persistent leukemia (>= 20% bone marrow cellularity and >= 5% bone marrow myeloblasts) proceed to remission induction course 2.

REMISSION INDUCTION COURSE 2: Patients receive bortezomib IV over 3-5 seconds on days 1 and 4; daunorubicin hydrochloride IV on days 1 and 2; and cytarabine IV continuously over 120 hours on days 1-5.

After completion of remission induction course 2, patients undergo bone marrow aspiration and biopsy for evaluation of response. Patients achieving a CR or PR proceed to remission consolidation therapy. Patients achieving a CRp proceed to remission consolidation therapy after platelet counts recover. Patients with residual leukemia who do not meet the criteria for PR are removed from the study.

REMISSION CONSOLIDATION THERAPY: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and intermediate-dose cytarabine IV over 3 hours on days 1-5. Patients then undergo bone marrow aspiration and biopsy for evaluation of response. Patients achieving a CR or who demonstrate continuing CR receive a second course of remission consolidation therapy beginning 2-4 weeks after blood counts recover.

After completion of study therapy, patients are followed every 2 months for 2 years, every 3 months for 2 years, and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocally histologically confirmed acute myeloid leukemia (AML)
* At least 20% blasts in the bone marrow based on WHO criteria
* No acute promyelocytic leukemia (M3)
* Antecedent hematologic disorder or myelodysplastic syndromes allowed provided the patient did not receive cytotoxic chemotherapy, including azacitidine and decitabine, for their pre-leukemic disorder
* Concurrent enrollment on CALGB-8461 required
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No ataxia, cranial neuropathy, or peripheral neuropathy >= grade 2
* LVEF >= 40% by ECHO or MUGA scan
* No signs or symptoms of congestive heart failure
* DLCO >= 50% (corrected for hemoglobin)
* No prior therapy for leukemia or pre-leukemic disorders, except for the following:

  * emergency leukapheresis;
  * emergency treatment for hyperleukocytosis with hydroxyurea;
  * cranial radiotherapy for CNS leukostasis (one dose only);
  * growth factor/cytokine support
* No other concurrent chemotherapy, except for the following:

  * I) steroids administered for adrenal failure, hypersensitivity reactions, or septic shock;
  * II) hormones administered for non-disease-related conditions (e.g., insulin for diabetes or estrogens or progestins for gynecologic indications)
* No concurrent palliative radiotherapy

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Attar, Principal Investigator — Cancer and Leukemia Group B
Locations (22):
- United States (22):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore-LIJ Health System CCOP, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Seffernick AE, Mrozek K, Nicolet D, Stone RM, Eisfeld AK, Byrd JC, Archer KJ. High-dimensional genomic feature selection with the ordered stereotype logit model. Brief Bioinform. 2022 Nov 19;23(6):bbac414. doi: 10.1093/bib/bbac414. PMID 36184192
- [Derived] Walker CJ, Kohlschmidt J, Eisfeld AK, Mrozek K, Liyanarachchi S, Song C, Nicolet D, Blachly JS, Bill M, Papaioannou D, Oakes CC, Giacopelli B, Genutis LK, Maharry SE, Orwick S, Archer KJ, Powell BL, Kolitz JE, Uy GL, Wang ES, Carroll AJ, Stone RM, Byrd JC, de la Chapelle A, Bloomfield CD. Genetic Characterization and Prognostic Relevance of Acquired Uniparental Disomies in Cytogenetically Normal Acute Myeloid Leukemia. Clin Cancer Res. 2019 Nov 1;25(21):6524-6531. doi: 10.1158/1078-0432.CCR-19-0725. Epub 2019 Aug 2. PMID 31375516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2008 and February 2010, 98 participants were recruited at 15 CALGB member institutions and their affiliated hospitals.
Pre-assignment Details: Three (3) participants did not begin treatment and were excluded from all analyses per study design
Groups:
- Bortezomib + Daunorubicin + Cytarabine: Bortezomib:
  Induction: 1.3 mg/sq m IV infusion Days 1,4,8,11 (Days 1, 4 only if 2nd induction)
  Consolidation: 0.7 OR 1 OR 1.3 mg/sq m IV infusion Days 1,4,8,11
  Cytarabine:
  Induction: 100 mg/sq m/day CIVI Days 1-7 (Days 1-5 only if 2nd induction) Consolidation: 2 g/sq m/day IV infusion Days 1-5
  Daunorubicin Induction: 60 mg/sq m IV infusion Days 1-3 (Days 1-2 if 2nd induction)
Period: Remission Induction
Arm/Group | Bortezomib + Daunorubicin + Cytarabine
Started | 95
Completed | 41
Not Completed | 54
Not completed — Progression | 6
Not completed — Failed induction | 8
Not completed — Adverse Event | 3
Not completed — Death | 10
Not completed — Refusal | 5
Not completed — Non protocol treatment | 17
Not completed — Other, not specified | 5
Period: Consolidation
Arm/Group | Bortezomib + Daunorubicin + Cytarabine
Started | 41
Completed | 20
Not Completed | 21
Not completed — Progression | 5
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Refused | 1
Not completed — Non protocol therapy | 13

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib + Daunorubicin + Cytarabine
Number analyzed (Participants) | 95
Age, Continuous [Median (Full Range); unit: years] | 67 [60 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 53
Region of Enrollment [Number; unit: participants]
  United States | 95
ECOG Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  participants
    0 - Fully Active | 31
    1 - Ambulatory, restricted strenuous activity | 55
    2 - Ambulatory, unable to perform work activities | 9

OUTCOME MEASURES:

1. Primary Outcome: Remission Induction Response
Description: Response was calculated according to Revised International Working Group (IWG) criteria for Acute myeloid leukemia (AML)
  A response was defined as the portion of participants who achieved a complete response (CR) or CR with incomplete platelet recovery(CRp) during induction.
  A CR is defined as those with > 20% cellularity of bone marrow biopsy, no presence of extramedullary leukemia for AML, <5 % myeloblast cells for bone marrow with peripheral blood and normal complete blood count (absolute neutrophils > 1000 mL and platelets >= 100,000 mL).
  A CRp is defined as a CR except platelets < 100,000 mL without need for transfusion.
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Bortezomib + Daunorubicin + Cytarabine
Number analyzed (Participants) | 95
participants
  Complete response | 62
  Complete response with incomplete platelet recover | 4

2. Primary Outcome: Participants Experiencing a Dose-limiting Toxicity (DLT) of Bortezomib When Administered in Combination With Intermediate-dose Cytarabine
Description: DLTs were considered only during the first cycle of consolidation therapy and included grade 3 or 4 sensory or autonomic neuropathy, persistent grade 4 thrombocytopenia or neutropenia at day 42 in the absence of AML,any grade 4 or 5 nonhematologic toxicity, and any grade 3 nonhematologic toxicity (excluding neuropathy and toxicities secondary to neutropenia and sepsis) that did not resolve to grade 2 by day 42 unless attributable to persistent or recurrent AML. Grade 4 anorexia (requiring total parenteral nutrition) and grade 4 fatigue (requiring bed rest) were not considered DLTs.
  Toxicity was graded per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Grading scale is as follows: grade 1: mild; grade 2: moderate; grade 3: Severe; grade 4: Life Threatening; grade 5: Death.
Time Frame: during consolidation cycle 1 (42 days)
Population: Participants who were registered to bortezomib consolidation were included in the analysis.
Measure: Number; unit: participants
Groups:
- Bortezomib (0.7 mg/m^2) + Int-DAC: Bortezomib (0.7 mg/m^2) + Intermediate Dose Cytarabine (Int-DAC)
- Bortezomib (1.0 mg/m^2) + Int-DAC: Bortezomib (1.0 mg/m^2) + Intermediate Dose Cytarabine (Int-DAC)
- Bortezomib (1.3 mg/m^2) + Int-DAC: Bortezomib (1.3 mg/m^2) + Intermediate Dose Cytarabine (Int-DAC)
Arm/Group | Bortezomib (0.7 mg/m^2) + Int-DAC | Bortezomib (1.0 mg/m^2) + Int-DAC | Bortezomib (1.3 mg/m^2) + Int-DAC
Number analyzed (Participants) | 3 | 3 | 17
participants | 0 | 0 | 1

3. Secondary Outcome: Disease-free Survival
Description: Disease-free survival (DFS) was measured as the interval from achievement of CR until relapse or death, regardless of cause. DFS was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 10 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib + Daunorubicin + Cytarabine
Number analyzed (Participants) | 95
months | 8 [6 to 12]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) as the interval from the on-study date until death. OS was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 10 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib + Daunorubicin + Cytarabine
Number analyzed (Participants) | 95
months | 12 [8 to 19]

ADVERSE EVENTS:
Groups:
- Bortezomib + Daunorubicin + Cytarabine: Induction: 60 mg/sq m IV infusion Days 1-3 (Days 1-2 if 2nd induction)
Arm/Group | Bortezomib + Daunorubicin + Cytarabine
Serious Adverse Events (participants affected / at risk) | 43/95
Other Adverse Events (participants affected / at risk) | 77/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib + Daunorubicin + Cytarabine (N=95)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 24 (27)
Hemoglobin (Blood and lymphatic system disorders) | 43 (51)
Hemolysis (e.g. immune hemolytic anemia drug-related hemolysis) (Blood and lymphatic system disorders) | 1 (1)
Lymphatics - Other (Specify __) (Blood and lymphatic system disorders) | 1 (1)
Cardiac Arrhythmia - Other (Specify __) (Cardiac disorders) | 13 (15)
Cardiac ischemia/infarction (Cardiac disorders) | 6 (6)
Cardiopulmonary arrest cause unknown (non-fatal) (Cardiac disorders) | 1 (1)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 16 (18)
Palpitations (Cardiac disorders) | 2 (2)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 8 (15)
Endocrine - Other (Specify __) (Endocrine disorders) | 1 (1)
Thyroid function high (hyperthyroidism thyrotoxicosis) (Endocrine disorders) | 1 (1)
Ocular/Visual - Other (Specify __) (Eye disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 36 (40)
Distension/bloating, abdominal (Gastrointestinal disorders) | 4 (4)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 (2)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 5 (5)
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (2)
Hemorrhage, GI (Gastrointestinal disorders) | 6 (6)
Ileus GI (functional obstruction of bowel i.e. neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 4 (5)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 30 (32)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 2 (2)
Ulcer GI (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (19)
Constitutional Symptoms - Other (Specify __) (General disorders) | 1 (1)
Death not associated with CTCAE term (General disorders) | 2 (2)
Edema: limb (General disorders) | 8 (8)
Edema: trunk/genital (General disorders) | 3 (3)
Edema:head and neck (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16 (17)
Fever (General disorders) | 1 (1)
Rigors/chills (General disorders) | 5 (5)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 29 (56)
Infection - Other (Specify __) (Infections and infestations) | 8 (8)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 10 (12)
Infection with unknown ANC (Infections and infestations) | 5 (5)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 2 (2)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 26 (29)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 29 (32)
Alkaline phosphatase (Investigations) | 10 (10)
Bilirubin (hyperbilirubinemia) (Investigations) | 25 (28)
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 5 (5)
Cardiac troponin I (cTnI) (Investigations) | 1 (1)
Creatinine (Investigations) | 8 (8)
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 2 (3)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 3 (3)
Leukocytes (total WBC) (Investigations) | 20 (24)
Lymphopenia (Investigations) | 16 (20)
Metabolic/Laboratory - Other (Specify __) (Investigations) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 43 (50)
PTT (Partial Thromboplastin Time) (Investigations) | 4 (4)
Platelets (Investigations) | 43 (51)
Prolonged QTc interval (Investigations) | 6 (6)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 3 (3)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 3 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 19 (20)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 10 (10)
Calcium serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 12 (12)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Glucose serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 13 (13)
Glucose serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 4 (4)
Magnesium serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 4 (4)
Phosphate serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 14 (14)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5 (5)
Potassium serum-low (hypokalemia) (Metabolism and nutrition disorders) | 19 (21)
Sodium serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 (2)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6 (6)
Uric acid serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 5 (5)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 8 (11)
CNS cerebrovascular ischemia (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 6 (7)
Hemorrhage CNS (Nervous system disorders) | 1 (1)
Neuropathy: cranial (Nervous system disorders) | 1 (2)
Neuropathy: motor (Nervous system disorders) | 3 (3)
Neuropathy: sensory (Nervous system disorders) | 16 (21)
Pain (Nervous system disorders) | 12 (30)
Somnolence/depressed level of consciousness (Nervous system disorders) | 7 (7)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 3 (3)
Taste alteration (dysgeusia) (Nervous system disorders) | 1 (1)
Vasovagal episode (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 5 (5)
Mood alteration (Psychiatric disorders) | 6 (7)
Personality/behavioral (Psychiatric disorders) | 1 (1)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 2 (2)
Glomerular filtration rate (Renal and urinary disorders) | 1 (1)
Hemorrhage GU (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 5 (5)
Renal/Genitourinary - Other (Specify __) (Renal and urinary disorders) | 3 (3)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Allergic rhinitis (including sneezing nasal stuffiness postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 19 (20)
Edema larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify __) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dermatology/Skin - Other (Specify __) (Skin and subcutaneous tissue disorders) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 22 (23)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (2)
Acute vascular leak syndrome (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (2)
Hemorrhage/Bleeding - Other (Specify __) (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (6)
Hypotension (Vascular disorders) | 26 (27)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Visceral arterial ischemia (non-myocardial) (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib + Daunorubicin + Cytarabine (N=95)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 50 (67)
Hemoglobin (Blood and lymphatic system disorders) | 76 (146)
Lymphatics - Other (Specify __) (Blood and lymphatic system disorders) | 3 (3)
Cardiac Arrhythmia - Other (Specify __) (Cardiac disorders) | 6 (7)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 12 (14)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 11 (12)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1)
Ocular surface disease (Eye disorders) | 1 (1)
Ocular/Visual - Other (Specify __) (Eye disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 10 (12)
Diarrhea (Gastrointestinal disorders) | 63 (86)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3 (3)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 3 (3)
Fistula, GI (Gastrointestinal disorders) | 2 (2)
Gastrointestinal - Other (Specify __) (Gastrointestinal disorders) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI (Gastrointestinal disorders) | 4 (5)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 12 (15)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 61 (95)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 2 (2)
Ulcer GI (Gastrointestinal disorders) | 1 (1)
Ulcer, GI (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 38 (49)
Edema: limb (General disorders) | 15 (18)
Edema: trunk/genital (General disorders) | 2 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 26 (36)
Fever (General disorders) | 3 (5)
Pain - Other (Specify, __) (General disorders) | 3 (3)
Rigors/chills (General disorders) | 16 (19)
Hepatobiliary/Pancreas - Other (Specify __) (Hepatobiliary disorders) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2)
Allergy/Immunology - Other (Specify __) (Immune system disorders) | 2 (3)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 46 (73)
Infection - Other (Specify __) (Infections and infestations) | 6 (7)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 6 (7)
Infection with unknown ANC (Infections and infestations) | 3 (3)
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 2 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 40 (65)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 49 (73)
Alkaline phosphatase (Investigations) | 16 (19)
Bilirubin (hyperbilirubinemia) (Investigations) | 34 (43)
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 10 (10)
Creatinine (Investigations) | 5 (7)
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 2 (4)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 4 (4)
Leukocytes (total WBC) (Investigations) | 23 (39)
Lymphopenia (Investigations) | 17 (28)
Metabolic/Laboratory - Other (Specify __) (Investigations) | 2 (2)
Neuroendocrine: ADH secretion abnormality (e.g. SIADH or low ADH) (Investigations) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 76 (142)
PTT (Partial Thromboplastin Time) (Investigations) | 8 (10)
Platelets (Investigations) | 75 (144)
Prolonged QTc interval (Investigations) | 2 (2)
Weight loss (Investigations) | 2 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 24 (30)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 22 (26)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 (1)
Calcium serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (3)
Calcium serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 26 (32)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 23 (39)
Glucose serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (2)
Magnesium serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5 (7)
Phosphate serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 21 (29)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5 (5)
Potassium serum-low (hypokalemia) (Metabolism and nutrition disorders) | 27 (36)
Sodium serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 (2)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 21 (29)
Uric acid serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 4 (4)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 7 (7)
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 12 (12)
Hemorrhage CNS (Nervous system disorders) | 1 (1)
Mental status (Nervous system disorders) | 1 (1)
Neurology - Other (Specify __) (Nervous system disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 3 (3)
Neuropathy: sensory (Nervous system disorders) | 21 (36)
Pain (Nervous system disorders) | 26 (70)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Taste alteration (dysgeusia) (Nervous system disorders) | 4 (5)
Tremor (Nervous system disorders) | 1 (1)
Vasovagal episode (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 9 (12)
Mood alteration (Psychiatric disorders) | 11 (16)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 2 (2)
Hemorrhage GU (Renal and urinary disorders) | 1 (1)
Obstruction, GU (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (including sneezing nasal stuffiness postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 14 (16)
Hemorrhage pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Hiccoughs (hiccups singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary/Upper Respiratory - Other (Specify __) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dermatology/Skin - Other (Specify __) (Skin and subcutaneous tissue disorders) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (4)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 (3)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 5 (6)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8 (9)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 53 (68)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 6 (6)
Urticaria (hives welts wheals) (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage/Bleeding - Other (Specify __) (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 16 (19)
Hypotension (Vascular disorders) | 28 (40)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Vascular - Other (Specify __) (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less